CLINICAL TRIAL: NCT01531218
Title: Randomized, Double-Blind, Placebo-Controlled Trial Of Azithromycin In Campylobacter Concisus Positive Patients With Diarrhea
Brief Title: Trial Of Azithromycin In Campylobacter Concisus Patients With Diarrhea
Acronym: Concisus2012
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aalborg University Hospital (Other); Slagelse Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT number: 2011-000808-18
Record Dates: First submitted 2012-02-08; First posted 2012-02-10 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-01

CONDITIONS: Diarrhea; Fever; Vomiting; Abdominal Pain
Keywords: Campylobacter; concisus; diarrhea; fever; abdominal pain; vomiting
MeSH Terms: conditions — Diarrhea; Fever; Vomiting; Abdominal Pain | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- azithromycin (Active Comparator): azithromycin 500mg
  Interventions: Drug: azithromycin
- placebo (Placebo Comparator): placebo 500mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: azithromycin — azithromycin, oral use, 500mg per day for 3 days in total. Total dose 1500mg
  Other Names: zitromax
  Arms: azithromycin
Drug: Placebo
  Arms: placebo

SUMMARY:
A randomized, double-blind, placebo-controlled clinical trial of azithromycin in Campylobacter concisus culture positive patients with diarrhea. The clinical characteristics of emerging Campylobacter concisus in adults is vomiting and persistent diarrhea. Whether patients may benefit from antibiotic treatment is unknown. The purpose of this trial is to investigate whether antibiotic treatment with azithromycin of Campylobacter concisus induced diarrhea can better the symptoms and shorten the duration of illness.

ELIGIBILITY:
Inclusion Criteria:

* Patients with culture-positive stool sample with Campylobacter concisus
* Diarrheic patients ≥ 18 years
* symptoms of diarrhea defined as three or more watery stools per day or
* two watery stools per day + at least one of the following symptoms: abdominal pain, nausea, vomiting or fever.
* Diarrheic symptoms for a minimum of 24 hours before enrollment.
* Diarrheic symptoms for a maximum of 21 days before enrollment.
* Informed oral and signed written consent, with documentation that all relevant information about the study is given to the patient.
* The patient must be willing and able to participate in the trial.

Exclusion Criteria:

* Hypersensitivity to azithromycin, erythromycin, macrolide or other ketolide-antibiotics
* Pregnancy or breastfeeding (if relevant).
* Culture positive stool sample with a Co-pathogen.
* Treatment with other antibiotics (in any stage 21 days before the first stool sample).
* Patients with severe liver disease.
* Patients with severe renal impairment (GFR <10 ml / min).
* Patients with congenital or documented acquired QT prolongation.
* Patients treated with other active drugs that prolong the QT interval such as: antiarrhythmics of classes IA and III, cisapride and terfenadine.
* Patients with electrolyte disorders, particularly hypokalemia and hypomagnesemia.
* Patients with clinically relevant bradycardia, arrhythmia or severe heart failure.
* Inflammatory bowel diseases
* Chronic diarrhea of known cause.
* Dementia.
* Serious illness less than 21 days from the planned entry into the study.
* Patients treated with medications that have interactions with azithromycin e.g. alkaloids, ciclosporin or amiodarone.
* Patients involved in the planning or execution of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Duration of diarrhea in days | up to 10 days

SECONDARY OUTCOMES:
number of stools/day | one day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Infectious Diseases, Aalborg Hospital, Aalborg, Denmark

REFERENCES:
- [Derived] Nielsen HL, Kirk KF, Bodilsen J, Ejlertsen T, Nielsen H. Azithromycin vs. Placebo for the Clinical Outcome in Campylobacter concisus Diarrhoea in Adults: A Randomized, Double-Blinded, Placebo-Controlled Clinical Trial. PLoS One. 2016 Nov 28;11(11):e0166395. doi: 10.1371/journal.pone.0166395. eCollection 2016. PMID 27893820